CLINICAL TRIAL: NCT05408962
Title: VeggieNutri - Nutritional and Metabolic Status of Vegetarian and Omnivorous Portuguese Adults
Brief Title: Nutritional and Metabolic Status of Vegetarian and Omnivorous Portuguese Adults
Acronym: VeggieNutri
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar De São João, E.P.E. (Other); Centro de Investigação em Tecnologias e Serviços de Saúde (Other); Rede de Investigação em Saúde (Other)
Responsible Party: Sponsor
Other Study IDs: VeggieNutri_2022
Record Dates: First submitted 2022-06-03; First posted 2022-06-07 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Diet, Vegetarian; Diet, Vegan; Nutritional Status; Metabolic Profile
Keywords: Vegetarian; Vegan; Diet quality; Metabolic profile; Nutritional status; Metabolic outcomes; Sustainable diets; Sustainability
MeSH Terms: interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples will be used to measure major metabolic outcomes. Urine samples will be used for oligoelement quantification (eg iodine).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- OMNI - omnivorous: Healthy omnivorous adults with ages between 18 and 65 years and having the reported dietary regimen for at least 1 year, free from any chronic condition such as metabolic, digestive, renal, haematological, endocrine or oncological diseases and presenting no food intolerances or eating disorders.
  Interventions: Other: Blood and urine collection, anthropometric analysis and answering to questionnaires
- LOV - lacto-ovovegetarians: Healthy lacto-ovovegetarians adults with ages between 18 and 65 years and having the reported dietary regimen for at least 1 year, free from any chronic condition such as metabolic, digestive, renal, haematological, endocrine or oncological diseases and presenting no food intolerances or eating disorders.
  Interventions: Other: Blood and urine collection, anthropometric analysis and answering to questionnaires
- VEG - vegan: Healthy vegan adults with ages between 18 and 65 years and having the reported dietary regimen for at least 1 year, free from any chronic condition such as metabolic, digestive, renal, haematological, endocrine or oncological diseases and presenting no food intolerances or eating disorders.
  Interventions: Other: Blood and urine collection, anthropometric analysis and answering to questionnaires

INTERVENTIONS:
Other: Blood and urine collection, anthropometric analysis and answering to questionnaires — During the visit to the recruitment center, participants will sign an informed consent. They will have to be in fasting condition for blood and urine collection. In addition they will answer the lifestyle questionnaire and the Food Frequency Questionnaire and will be submitted to an anthropometric analysis and evaluation of blood preassure and heart rate.

SUMMARY:
Vegetarian diets have low environmental footprints and are potential solutions to address climate change and the 2030 Agenda on the Sustainable Development Goals. Currently, there is no information regarding the nutritional quality of vegetarian diets in Portugal. As the trend for vegetarianism increases in the country, the aim of this study is to examine and compare nutritional and metabolic outcomes among vegetarian and non-vegetarian populations. We aim to implement a cross-sectional study that includes a total of 400 (distributed among the three diferent groups of omnivorous, lacto-ovovegatarians and vegans) healthy Portuguese adults aged 18-64 years. Blood and urine samples will be collected. Participants will be assessed for blood pressure, anthropometric parameters, micronutrient status, blood lipids, glicaemia and insuline resistance and will complete a validated food frequency questionnaire as well as a sociodemographic and lifestyle questionnaire. Dietary and nutrient analysis will be conducted to assess diet quality and nutritional inadequacies. The current proposal provides an unique opportunity to characterize and compare different population groups clustered by dietary behaviour and provide evidence that help achieve healthy and sustainable diets in Portugal.

DETAILED DESCRIPTION:
Plant-based diets have been proven to be sustainable and to have low environmental impact, highlighting the importance of promoting a dietary shift towards plant-based diets, with reduction in the consumption of animal food sources. In particular, vegetarian diets can refer to vegan (VEG) diets that completely exclude all animal derived foods or to lacto-ovo vegetarians (LOV) which include eggs and milk products and have low environmental footprint compared with omnivorous dietary patterns. Vegetarian diets are gaining popularity around the world. The reasons to follow a vegetarian diet are diverse and reported to be related to religion, animal welfare, sustainability and environmental reasons, as well as health related concerns. Literature has shown several health benefits of these diets. Regarding the efficiency of vegetarianism in promoting weight loss, studies in which a lacto-ovo vegetarian or vegan diet are administered to participants show that participants with previous plant based-diets that do not fully adhere to the prescribed weight loss diet loose more weight when compared to non-vegetarians. Moreover, vegan diets have been shown to be more effective in improving body composition and insulin resistance, when compared to an omnivorous diet. Despite the above referred evidence regarding beneficial effects on weight loss, some studies find no statistical differences on weight loss promoted by vegetarians, omnivorous or Mediterranean diets. Plant-based diets were also found to improve glycaemic control and insulin sensitivity. In fact, there is evidence on vegetarians having lower fasting insulin level and higher insulin sensitivity compared with matched omnivores. Moreover, these diets are considered to have a low inflammatory load to the point of being considered as an approach to lower inflammatory markers in patients with coronary artery disease. Nevertheless, since vegetarian diets are restrictive, they may give rise to nutritionally unbalanced regimens, particularly when adopted without nutritional counselling. In fact, several studies link vegetarian diets to poor nutritional status, including micronutrient deficiency. In this context, the great rise of vegetarian habits among Portuguese population, which are reported to have quadruplicated in the last 10 years, poses important health concerns. Nevertheless, data on the nutritional status characteristics and metabolic profile of such consumers and of the nutritional adequacy of their diet are scarce, particularly comparing with people with omnivorous dietary regimens.

So, it is crucial to assess the quality of vegetarian diets in the country, identifying clear health benefits and risks from a nutritional perspective. Considering the importance of promoting environmentally sustainable diets at national level and the lack of data regarding the diet quality of vegetarian diets in the country, we propose the implementation of the first cross-sectional study in the country to investigate and compare nutritional and health parameters among vegetarian and omnivorous populations. The current proposal provides an unique opportunity to characterize and compare different population groups clustered by dietary behaviour and identify potential risks and gaps to attain health and environmental goals, such as contributing to the Portugal commitments to achieve the 2030 Agenda on the Sustainable Development Goals.

ELIGIBILITY:
Inclusion Criteria:

* being a healthy adult
* being aged between 18 and 65 years
* having the reported dietary regimen for at least 1 year

Exclusion Criteria:

* being free from metabolic disorders
* being free from digestive disorders
* being free from renal disorders
* being free from haematological disorders
* being free from endocrine disorders
* being free from oncological diseases
* being free from food intolerances
* being free from eating disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from general population. During advertisement, people will be invited to express their interest by filling in an online form which will include information about participation eligibility (eligibility criteria explained bellow). On recruitment day eligible participants will be asked to visit the recruitment center in fasting for blood and urine collection. In addition they will sign an informed consent, answer the lifestyle questionnaire and the Food Frequency Questionnaire and will be submitted to an anthropometric analysis and evaluation of blood preassure and heart rate.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Diet Quality Index for each regimen | 7 months
  Diet quality will be assessed through a Diet Quality Index (DQI) created by VeggieNutri's workteam. DQI is a tool that quantifies the quality of an individual's intake, scoring their food intake, assessed buy a Food Frequency Questionnaire (FFQ). Each question regarding their food intake will be scored from 0 to 10 points, depending on how close they are to complying with guidelines and recommendations (the closer to complying, the highest the scoring and the farthest, the lower the scoring).
Nutritional inadequacy prevalences | 11 months
  Nutritional inadequacy prevalences will be calculated based on DQI scores and also on reference values for micronutrients in blood or urine.

SECONDARY OUTCOMES:
Levels of vitamins B12, B6, B9 and D, homocysteine, iron, selenium, calcium, zinc and magnesium | 6 months
  Measured in blood samples.
Waist circunference and percentage of body fat | 6 months
  Assessed through anthropometric analysis including bioelectrical impedance, on the recruitment day.
Fasting glycaemia and HOMA-IR | 6 months
  Quantification of fasting blood glucose and insulin.
Blood LDL, HDL and total cholesterol and triglycerides | 6 months
  Assessed through the analysis of blood samples.
Urinary iodine concentration | 6 months
  Assessed through the analysis of urine samples.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Keating, PhD, Principal Investigator — Universidade do Porto
Locations (1):
- Faculty of Medicine (FMUP), Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided